CLINICAL TRIAL: NCT03286166
Title: A Randomized Controlled Trial to Evaluate the Efficiency of Serum Tears Made With Genius PRP for Improving Signs and Symptoms in Dry Eye Disease (DED)
Brief Title: Single Center, Prospective, Randomized, Controlled, Non-significant Risk
Status: Withdrawn | Type: Observational
Why Stopped: due to funding issues
Sponsor: Toyos Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: TOYOS-GENIUSPRP-17-01
Record Dates: First submitted 2017-09-07; First posted 2017-09-18 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study arm: 20 subjects will undergo one session of PRP in which 60 cc of blood is drawn and centrifuged into 3 months of autologous serum tears.
  • Subjects will utilize autologous tears twice daily in the study eye.
- Control Arm: Subjects in the control arm will receive study vehicle to be used twice daily in the left eye.

SUMMARY:
A randomized controlled trial to evaluate the efficiency of serum tears made with Genius PRP for improving signs and symptoms in Dry Eye Disease (DED).

Single center, Prospective, Randomized, Controlled, Non-significant risk

DETAILED DESCRIPTION:
Genius PRP is a class II medical device with an 510(k)FDA clearance for platelet and plasma separation for bone graft handling.

Subjects will sign the IC form within one week of being having been provided the form, at which time they will undergo the following assessments:

* Routine ophthalmology tests (biomicroscopy, BCVA and IOP) including corneal fluorescein staining and lissamine green conjunctival staining
* Measurement of tear break up time (TBUT) in both eyes. These values will be used as baseline.
* Self-administration of the Eye Dryness Scale; 0-100 visual analogue scale. This score will be used as baseline.
* Self-administration of Visual Analog Pain Scale
* Eligible subjects will be randomized with right eye to receive PRP and left eye to receive vehicle eye drops in the same dosage.

Outcome measures will be assessed in both eyes.

ELIGIBILITY:
Inclusion Criteria:

* 1) Able to read, understand and sign an Informed Consent (IC) form 2) 22-85 years of age 3) Able and willing to comply with the treatment/follow-up schedule and requirements 4) Tear break up time of less than 10 seconds in both eyes 5) SPK in the conjunctiva and/or cornea of each eye 6) Eye dryness scale of 40 or greater at baseline for each eye 7) Self- reported ocular pain from dry eye disease

Exclusion Criteria:

1) Unwilling to discontinue use of contact lenses for the duration of the study 2) Ocular surgery or eyelid surgery, within 3 months prior to screening 3) Neuro-paralysis in the planned treatment area, within 6 months prior to screening 4) Other uncontrolled eye disorders affecting the ocular surface, for example active allergies 5) Punctal plugs placed within past 90 days 6) Pre-cancerous lesions, skin cancer or pigmented lesions in the planned treatment area 7) Uncontrolled infections or uncontrolled immunosuppressive diseases 8) Subjects with current ocular infections. 9) New prescription eye drops for dry eye or glaucoma or omega 3 supplements prescribed within 90 days prior to screening, excluding artificial tears 10) New topical treatments within the area to be treated, or oral therapies, within 3 months prior to screening- except over-the-counter acetaminophen-based analgesics for pain management 11) Change in dosage of any systemic medication, within 3 months prior to screening 12) Anticipated relocation or extensive travel outside of the local study area preventing compliance with follow-up over the study period 13) Legally blind in one or both eyes 14) First IPL treatment, within 3 months prior to screening 15) Any condition revealed during the eligibility screening process whereby the investigator deems the subject inappropriate for this study

-

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 20 male or female subjects, aged 22-85, with signs and symptoms of DED and ocular pain related to DED in the opinion of the investigator
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The difference in the change of EDS score from baseline and the tear breakup time from baseline to follow-up, between study eyes in the study arm and study eyes in the control arm | 3 months
  * Change in EDS questionnaire from baseline
  * Change in TBUT from baseline.

SECONDARY OUTCOMES:
The improvement of signs and visual analog pain scale in the study group is larger than the improvement of signs in the control group | 3 months
  * Change in corneal and/or conjunctival SPK
  * Visual analog pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Toyos Clinic, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No